CLINICAL TRIAL: NCT01526551
Title: A Study to Compare the Impact of a School Based HPV Vaccination Program on Vaccination Uptake and Completion Rates Among High School Students in Rural, Southeastern Kentucky
Brief Title: A Study to Compare the Impact of a School Based HPV Program on Vaccination Uptake and Completion Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Cumberland District Health Department (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LCDHD-12-HPV
Record Dates: First submitted 2011-12-22; First posted 2012-02-06 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Human Papillomavirus
Keywords: Human Papillomavirus
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Schools (Experimental): High school students attending Wayne County and Monticello Ind. schools will be given opportunity to receive HPV Vaccine and HPV-related Health Education and Reduction of barriers to being vaccinated.
  Interventions: Other: HPV Vaccine and HPV-related Health Education; Other: Reduction of barriers

INTERVENTIONS:
Other: HPV Vaccine and HPV-related Health Education — Increased education of HPV-related diseases and HPV vaccine
Other: Reduction of barriers — Eliminate structural and financial barriers to being vaccinated
  Other Names: School based delivery of HPV vaccine

SUMMARY:
The purpose of this study is to evaluate the impact of a school-based Human Papillomavirus (HPV) vaccination program to determine if the combination of increased disease and vaccine education coupled with the removal of barriers will positively impact the HPV vaccination uptake and completion rates among students.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of a school-based HPV vaccination program. The intervention will consists of: provision of HPV vaccine information and consent forms for parents delivered in the back-to-school packets; school-nurse delivered student education; removal of barriers (scheduling, transportation and parental presence); changing of social norms; and the provision of free HPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Must have not completed three dose series of HPV vaccine
* Must be a student at Wayne County or Monticello High School in KY

Exclusion Criteria:

* Completed three dose series
* Pregnant
* Contraindication to vaccine ingredients

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 935 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Weyman, M.D., Principal Investigator — Lake Cumberland District Health Department
Locations (2):
- United States (2):
  - Monticello High School, Monticello, Kentucky
  - Wayne County High School, Monticello, Kentucky

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention School: High school students attending Wayne County and Monticello Ind. schools will be given opportunity to receive HPV vaccination in school clinic
  HPV Vaccine and Disease Education: Increased education of disease and vaccine
  Reduction of barriers: eliminate barriers to being vaccinated
Period: Overall Study
Arm/Group | Intervention School
Started | 935
Completed | 511
Not Completed | 424
Not completed — Lack of returned parental consent form | 424

BASELINE CHARACTERISTICS:
Arm/Group | Intervention School
Number analyzed (Participants) | 511
Age, Customized [Number; unit: participants]
  Ages 12-20 | 511
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240
  Male | 271
Grade [Number; unit: participants]
  9th grade | 142
  10th grade | 128
  11th grade | 116
  12th grade | 124
  missing | 1
Insurance Status [Number; unit: participants]
  Insured | 114
  Medicaid/KCHIP | 182
  No Insurance | 22
  Underinsured | 28
  Unknown | 165
Prior doses (baseline) [Number; unit: participants]
  0 | 447
  1 | 9
  2 | 5
  3 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Students Who Initiated the HPV Vaccine Series as a Result of the School-based Program
Description: Number of students who returned a parental consent form and ultimately initiated the HPV vaccine series as a result of the school-based program
Time Frame: August 2012-June 2013
Measure: Number; unit: participants
Arm/Group | Intervention School
Number analyzed (Participants) | 511
participants | 315

2. Primary Outcome: Number of Students Who Completed HPV Vaccination as a Result of the School-based Program
Description: Number of students who returned a parental consent form and ultimately completed the full HPV vaccination series as a result of the school-based program
Time Frame: August 2012 -- June 2013
Measure: Number; unit: participants
Arm/Group | Intervention School
Number analyzed (Participants) | 511
participants | 288

ADVERSE EVENTS:
Time Frame: August 2012-June 2013
Description: Staff developed and implemented a protocol that allowed for documentation of adverse vaccine reactions among all vaccine-receiving students.
Arm/Group | Intervention School
Serious Adverse Events (participants affected / at risk) | 0/511
Other Adverse Events (participants affected / at risk) | 0/511

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No